CLINICAL TRIAL: NCT01889173
Title: A Single-Dose, Open-Label, Randomized, Parallel-Design Study Of The Comparative Pharmacokinetics And Safety Of TNX-102 2.8 mg SL Tablets (With Potassium Phosphate) At 2.8 mg, TNX-102-B 2.8 mg SL Tablets (With Sodium Phosphate) At 2.8 mg, TNX-102-C 2.8 mg SL Tablets (With Trisodium Citrate) At 2.8 mg, And Cyclobenzaprine 5 mg Oral Tablets In Healthy Adults
Brief Title: Comparative Pharmacokinetics and Safety of 3 Different Formulations of TNX-102 2.8 mg SL Tablets and Cyclobenzaprine 5 mg Oral Tablet in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CY-F104
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Adults
MeSH Terms: interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TNX-102 SL Tablets at 2.8 mg (Experimental): 1 x TNX-102 SL Tablets (with potassium phosphate) at 2.8 mg
  Interventions: Drug: TNX-102 SL Tablets at 2.8 mg
- TNX-102-B SL Tablets at 2.8 mg (Experimental): 1 x TNX-102-B SL Tablets (with sodium phosphate) at 2.8 mg
  Interventions: Drug: TNX-102-B SL Tablets at 2.8 mg
- TNX-102-C SL Tablets at 2.8 mg (Experimental): 1 x TNX-102-C SL Tablets (with trisodium citrate) at 2.8 mg
  Interventions: Drug: TNX-102-C SL Tablets at 2.8 mg
- Cyclobenzaprine tablets (Active Comparator): 1 x 5 mg cyclobenzaprine oral tablet
  Interventions: Drug: Cyclobenzaprine tablets

INTERVENTIONS:
Drug: TNX-102 SL Tablets at 2.8 mg — 1 x TNX-102 SL Tablet (with potassium phosphate) at 2.8 mg held under the tongue until dissolution, without swallowing or chewing it.
  Arms: TNX-102 SL Tablets at 2.8 mg
Drug: TNX-102-B SL Tablets at 2.8 mg — 1 x TNX-102-B SL Tablet (with sodium phosphate) at 2.8 mg held under the tongue until dissolution, without swallowing or chewing it.
  Arms: TNX-102-B SL Tablets at 2.8 mg
Drug: TNX-102-C SL Tablets at 2.8 mg — 1 x TNX-102-C SL Tablet (with trisodium citrate) at 2.8 mg held under the tongue until dissolution, without swallowing or chewing it.
  Arms: TNX-102-C SL Tablets at 2.8 mg
Drug: Cyclobenzaprine tablets — 1 x 5 mg cyclobenzaprine tablet, swallowed with 240 mL of room-temperature water
  Arms: Cyclobenzaprine tablets

SUMMARY:
Very low dose (VLD) cyclobenzaprine at bedtime has shown promise as a treatment for fibromyalgia, but the chemistry of cyclobenzaprine requires new formulation technology for bedtime use. The present trial is designed to assess the safety and tolerability of 3 different formulations of TNX-102 2.8 mg SL Tablets (a new formulation of cyclobenzaprine designed to result in increased dosage precision and decreased potential for morning grogginess) and to compare the bio-availability of 3 different formulations of TNX-102 2.8 mg SL Tablets (TNX-102 with potassium phosphate, TNX-102-B with sodium phosphate, and TNX-102-C with trisodium citrate) to that of cyclobenzaprine (5 mg tablets).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Male or female
* 18-65 years old
* Non-smoker
* BMI > 18.5 and < 30.0
* With medically acceptable form of contraception (female only)
* With signed informed consent

Exclusion Criteria:

* Any clinically significant abnormality including ECG abnormalities or vital sign abnormalities (systolic blood pressure < 90 or > 140 mmHg,
* Diastolic blood pressure lower < 50 or > 90 mmHg, or heart rate < 50 or > 100 BPM)
* Any abnormal laboratory test (including positivity for Hep B, Hep C, HIV, and
* Hemoglobin < 128 g/L (males) or < 115 g/L (females) and hematocrit < 0.37 L/L (males) or < 0.32 L/L (females))
* History of alcohol or drug abuse or dependence within 1 year and/or positive drug, cotinine, or alcohol tests
* Use of any drug (within 30 days), supplement, or food (within 14 days) known to induce or inhibit hepatic drug metabolism prior to study medication
* Positive pregnancy test, breastfeeding or lactating
* Use of medication other than hormonal contraceptives or topical products, including OTC, natural health products, MAO inhibitors
* Participation in an investigational study within 30 days prior to dosing
* Donation of plasma (within 7 days), or donation or loss of blood of 50-499 mL (within 30 days), or of > 499 mL (within 56 days) prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Measured levels of cyclobenzaprine and norcyclobenzaprine in plasma and urine | 26 time points per period for blood assessment ; 2 pooled analyses in urine.
  Blood samples will be taken per period: within 30 minutes pre-dose and 2, 3.5, 5, 10, 20, 30, and 45 minutes and 1, 2, 2.5, 3, 3.33, 3.67, 4, 4.33, 4.67, 5, 5.5, 6, 8, 12, 16, 24, 36, and 48 hours post-dose. A single urine sample will be collected within 30 minutes pre-dose (one sample), and urine will be pooled from 0-24 and 24-48 hours post-dose.
Safety and tolerability of the 3 formulations of TNX-102 SL Tablets at 2.8 mg | Continuously until the end (day 3) of the study period + Telephone follow-up 7-13 days after dosing (total duration: about 1 month)
  Every adverse events occurring during the study period will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Seth M. Lederman, MD, Study Chair — Tonix Pharmaceuticals, Inc.; Jeffrey P. Kitrelle, MD, Study Director — Tonix Pharmaceuticals, Inc.; Denis Audet, MD, Principal Investigator — PharmaNet
Locations (1):
- PharmaNet, Inc., Québec, Quebec, Canada